CLINICAL TRIAL: NCT06002841
Title: Extracellular Vesicles From Mesenchymal Cells in the Treatment of Acute Respiratory Failure Associated With SARS-CoV-2 and Other Etiologies: a Clinical Trial, Randomized, Double-blind.
Brief Title: Extracellular Vesicles From Mesenchymal Cells in the Treatment of Acute Respiratory Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Hospital Sao Rafael (Other); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVs_2023
Record Dates: First submitted 2023-07-27; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Severe Acute Respiratory Syndrome (SARS); Acute Respiratory Distress Syndrome (ARDS); Pneumonia
Keywords: SARS-CoV-2; intravenous therapy; extracellular vesicles; ARDS; mesenchymal cells
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome; Pneumonia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: The treatment and placebo solutions will be indistinguishable in terms of their appearance. Stringent protocols will be established to guarantee that the physicians responsible for assessing patient safety, evaluating efficacy outcomes, and conducting laboratory analyses will be blinded to the randomization codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV group (Experimental): will consist of 10 participants who will receive two infusions of 25 mL of the investigational product (Plasma-Lyte A solution containing EVs obtained from MSCs), intravenously, at intervals of 48 h.
  Interventions: Biological: intravenous treatment with EVs
- Placebo group (Placebo Comparator): will consist of 5 participants who will receive an equal volume of Plasma-Lyte A, intravenously, following the same schedule as the IV group: two infusions with an interval of 48 hours.
  Interventions: Biological: intravenous treatment with placebo solution

INTERVENTIONS:
Biological: intravenous treatment with EVs — intravenous treatment with extracellular vesicles
  Arms: EV group
Biological: intravenous treatment with placebo solution — intravenous treatment with placebo solution (without extracellular vesicles)
  Arms: Placebo group

SUMMARY:
This is a phase I/II, randomized, double-blind, placebo-controlled clinical trial that will evaluate the safety and potential efficacy of therapy with extracellular vesicles (EVs) obtained from mesenchymal stromal cells (MSCs), patients with moderate to severe acute respiratory distress syndrome due to COVID-19 or other etiology. Participants will be allocated to receive EVs obtained from MSCs or placebo (equal volume of Plasma-Lyte A). Blinding will cover the participants, the multidisciplinary intensive care team and the investigators.

DETAILED DESCRIPTION:
The studied population will consist of 15 patients diagnosed with acute respiratory failure syndrome admitted to the intensive care unit of Hospital São Rafael. This research aims to assess the safety and potential effectiveness of intravenous therapy using extracellular vesicles derived from mesenchymal cells in patients with moderate to severe acute respiratory distress syndrome. The treatment group will receive intravenous administration of extracellular vesicles obtained from mesenchymal cells, while the control group will receive a placebo.

EV group: will consist of 10 participants who will receive two infusions of 25 mL of the investigational product (Plasma-Lyte A solution containing EVs obtained from MSCs), intravenously, at intervals of 48 h.

Placebo group: will consist of 5 participants who will receive an equal volume of Plasma-Lyte A, intravenously, following the same schedule as the IV group: two infusions with an interval of 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old;
* Chest CT radiological image with ground-glass opacities or chest X-ray with - bilateral infiltrates characteristic of pulmonary edema;
* In invasive mechanical ventilation with PEEP 5 cm H2O and PaO2/FiO2<250mmHg;
* Respiratory failure not explained by cardiac causes or fluid overload.

Exclusion Criteria:

* Unable to provide informed consent;
* Pregnancy or breastfeeding;
* Patients with active malignancy who have received chemotherapy in the last 2 years;
* Life expectancy of less than 6 months or in exclusive palliative care;
* Severe liver failure, with a Child-Pugh score > 12;
* Previous renal failure: patients already undergoing dialysis or patients with GFR < 30ml/min/1.73 m2
* Clinical or radiological suspicion of tuberculosis;
* Chronic respiratory failure;
* Use of ECMO;
* Moribund (high probability of death within the next 48 hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Measure administration of extracellular vesicles (EVs) up to 28 days | 28 days
  Measure as reported adverse events up to 28 days after treatment or placebo administration to evaluate safety of treatment

SECONDARY OUTCOMES:
All-cause mortality | Day 14 and day 28
  at days 14 and 28 after randomization;
Variation in the Ratio PaO2/FiO2 | Baseline, day 01, day 02 and day 07
  PaO2 (arterial partial pressure of oxygen)/FiO2 (fraction of inspired oxygen) on the day of randomization and at 24 hours, 48 hours and 7 days after the first infusion;
Variation in the SOFA index | day 01, day 02, day 07, day 09, day 14 and day 29
  Variation in the SOFA index (Assessment of Sequential Organ Failure) at the time of randomization and during follow-up until discharge from the intensive care unit;
Exploratory laboratory analysis | 30 days
  variation in total and differential laboratory analysis.
Duration of the period of hospitalization | 30 days
  from hospital time in the intensive care unit (ICU)
Duration of the period of ICU ventilation | 30 days
  If applicable,will be measured the time of mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Souza, M.D, Principal Investigator — Instituto D'Or de Pesquisa e Ensino (IDOR), Salvador, Brazil; Patrícia Rocco, M.D, Principal Investigator — Universidade Federal do Rio de Janeiro (UFRJ)
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abels ER, Breakefield XO. Introduction to Extracellular Vesicles: Biogenesis, RNA Cargo Selection, Content, Release, and Uptake. Cell Mol Neurobiol. 2016 Apr;36(3):301-12. doi: 10.1007/s10571-016-0366-z. Epub 2016 Apr 6. PMID 27053351
- [Background] Alipoor SD, Mortaz E, Garssen J, Movassaghi M, Mirsaeidi M, Adcock IM. Exosomes and Exosomal miRNA in Respiratory Diseases. Mediators Inflamm. 2016;2016:5628404. doi: 10.1155/2016/5628404. Epub 2016 Sep 25. PMID 27738390
- [Background] Antunes MA, Braga CL, Oliveira TB, Kitoko JZ, Castro LL, Xisto DG, Coelho MS, Rocha N, Silva-Aguiar RP, Caruso-Neves C, Martins EG, Carvalho CF, Galina A, Weiss DJ, Lapa E Silva JR, Lopes-Pacheco M, Cruz FF, Rocco PRM. Mesenchymal Stromal Cells From Emphysematous Donors and Their Extracellular Vesicles Are Unable to Reverse Cardiorespiratory Dysfunction in Experimental Severe Emphysema. Front Cell Dev Biol. 2021 May 31;9:661385. doi: 10.3389/fcell.2021.661385. eCollection 2021. PMID 34136481
- [Background] de Castro LL, Xisto DG, Kitoko JZ, Cruz FF, Olsen PC, Redondo PAG, Ferreira TPT, Weiss DJ, Martins MA, Morales MM, Rocco PRM. Human adipose tissue mesenchymal stromal cells and their extracellular vesicles act differentially on lung mechanics and inflammation in experimental allergic asthma. Stem Cell Res Ther. 2017 Jun 24;8(1):151. doi: 10.1186/s13287-017-0600-8. PMID 28646903
- [Background] Cruz FF, Borg ZD, Goodwin M, Sokocevic D, Wagner DE, Coffey A, Antunes M, Robinson KL, Mitsialis SA, Kourembanas S, Thane K, Hoffman AM, McKenna DH, Rocco PR, Weiss DJ. Systemic Administration of Human Bone Marrow-Derived Mesenchymal Stromal Cell Extracellular Vesicles Ameliorates Aspergillus Hyphal Extract-Induced Allergic Airway Inflammation in Immunocompetent Mice. Stem Cells Transl Med. 2015 Nov;4(11):1302-16. doi: 10.5966/sctm.2014-0280. Epub 2015 Sep 16. PMID 26378259
- [Background] De Jong OG, Van Balkom BW, Schiffelers RM, Bouten CV, Verhaar MC. Extracellular vesicles: potential roles in regenerative medicine. Front Immunol. 2014 Dec 3;5:608. doi: 10.3389/fimmu.2014.00608. eCollection 2014. PMID 25520717
- [Background] Kordelas L, Rebmann V, Ludwig AK, Radtke S, Ruesing J, Doeppner TR, Epple M, Horn PA, Beelen DW, Giebel B. MSC-derived exosomes: a novel tool to treat therapy-refractory graft-versus-host disease. Leukemia. 2014 Apr;28(4):970-3. doi: 10.1038/leu.2014.41. No abstract available. PMID 24445866
- [Background] Lanyu Z, Feilong H. Emerging role of extracellular vesicles in lung injury and inflammation. Biomed Pharmacother. 2019 May;113:108748. doi: 10.1016/j.biopha.2019.108748. Epub 2019 Mar 14. PMID 30877881
- [Background] Lasser C, Jang SC, Lotvall J. Subpopulations of extracellular vesicles and their therapeutic potential. Mol Aspects Med. 2018 Apr;60:1-14. doi: 10.1016/j.mam.2018.02.002. Epub 2018 Feb 16. PMID 29432782
- [Background] Naji A, Eitoku M, Favier B, Deschaseaux F, Rouas-Freiss N, Suganuma N. Biological functions of mesenchymal stem cells and clinical implications. Cell Mol Life Sci. 2019 Sep;76(17):3323-3348. doi: 10.1007/s00018-019-03125-1. Epub 2019 May 4. PMID 31055643
- [Background] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Background] Sengupta V, Sengupta S, Lazo A, Woods P, Nolan A, Bremer N. Exosomes Derived from Bone Marrow Mesenchymal Stem Cells as Treatment for Severe COVID-19. Stem Cells Dev. 2020 Jun 15;29(12):747-754. doi: 10.1089/scd.2020.0080. Epub 2020 May 12. PMID 32380908
- [Background] Silva JD, de Castro LL, Braga CL, Oliveira GP, Trivelin SA, Barbosa-Junior CM, Morales MM, Dos Santos CC, Weiss DJ, Lopes-Pacheco M, Cruz FF, Rocco PRM. Mesenchymal Stromal Cells Are More Effective Than Their Extracellular Vesicles at Reducing Lung Injury Regardless of Acute Respiratory Distress Syndrome Etiology. Stem Cells Int. 2019 Aug 21;2019:8262849. doi: 10.1155/2019/8262849. eCollection 2019. PMID 31531026
- [Background] Shi MM, Yang QY, Monsel A, Yan JY, Dai CX, Zhao JY, Shi GC, Zhou M, Zhu XM, Li SK, Li P, Wang J, Li M, Lei JG, Xu D, Zhu YG, Qu JM. Preclinical efficacy and clinical safety of clinical-grade nebulized allogenic adipose mesenchymal stromal cells-derived extracellular vesicles. J Extracell Vesicles. 2021 Aug;10(10):e12134. doi: 10.1002/jev2.12134. Epub 2021 Aug 14. PMID 34429860
- [Background] D'Souza-Schorey C, Schorey JS. Regulation and mechanisms of extracellular vesicle biogenesis and secretion. Essays Biochem. 2018 May 15;62(2):125-133. doi: 10.1042/EBC20170078. Print 2018 May 15. PMID 29666210
- [Background] Tieu A, Lalu MM, Slobodian M, Gnyra C, Fergusson DA, Montroy J, Burger D, Stewart DJ, Allan DS. An Analysis of Mesenchymal Stem Cell-Derived Extracellular Vesicles for Preclinical Use. ACS Nano. 2020 Aug 25;14(8):9728-9743. doi: 10.1021/acsnano.0c01363. Epub 2020 Aug 4. PMID 32697573
- [Background] Wiklander OP, Nordin JZ, O'Loughlin A, Gustafsson Y, Corso G, Mager I, Vader P, Lee Y, Sork H, Seow Y, Heldring N, Alvarez-Erviti L, Smith CI, Le Blanc K, Macchiarini P, Jungebluth P, Wood MJ, Andaloussi SE. Extracellular vesicle in vivo biodistribution is determined by cell source, route of administration and targeting. J Extracell Vesicles. 2015 Apr 20;4:26316. doi: 10.3402/jev.v4.26316. eCollection 2015. PMID 25899407
- [Background] Zhou T, He C, Lai P, Yang Z, Liu Y, Xu H, Lin X, Ni B, Ju R, Yi W, Liang L, Pei D, Egwuagu CE, Liu X. miR-204-containing exosomes ameliorate GVHD-associated dry eye disease. Sci Adv. 2022 Jan 14;8(2):eabj9617. doi: 10.1126/sciadv.abj9617. Epub 2022 Jan 12. PMID 35020440
- [Background] Zhu YG, Feng XM, Abbott J, Fang XH, Hao Q, Monsel A, Qu JM, Matthay MA, Lee JW. Human mesenchymal stem cell microvesicles for treatment of Escherichia coli endotoxin-induced acute lung injury in mice. Stem Cells. 2014 Jan;32(1):116-25. doi: 10.1002/stem.1504. PMID 23939814